CLINICAL TRIAL: NCT06850623
Title: A Phase 2 Study to Investigate the Efficacy and Safety of Acoustic Cluster Therapy With Modified FOLFIRINOX in Patients With Locally Advanced Pancreatic Cancer
Brief Title: Acoustic Cluster Therapy (ACT) With Chemotherapy for the Treatment of Locally Advanced Pancreatic Cancer
Acronym: ENACT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EXACT Therapeutics AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EX-2-P2-2023
Record Dates: First submitted 2025-01-15; First posted 2025-02-27 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma
Keywords: pancreatic cancer; PS101; ultrasound; microbubbles; Pancreatic Ductal Carcinoma; locally advanced pancreatic cancer; first line treatment; chemotherapy; Acoustic Cluster Therapy; mFOLFIRINOX
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Pancreatic Ductal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Acoustic Cluster Therapy (ACT) with mFOLFIRINOX (Experimental)
  Interventions: Combination Product: Acoustic Cluster Therapy; Drug: Modified FOLFIRINOX

INTERVENTIONS:
Combination Product: Acoustic Cluster Therapy — Drug: PS101; Device: Ultrasound
Drug: Modified FOLFIRINOX — Chemotherapy

SUMMARY:
The purpose of the study is to assess the efficacy and safety of Acoustic Cluster Therapy (ACT) when given in addition to chemotherapy for treatment of Locally Advanced Pancreatic Cancer.

DETAILED DESCRIPTION:
Patients with Locally Advanced Pancreatic Cancer who have not received prior treatment to their pancreatic cancer will receive ACT treatment (the drug PS101 and ultrasound application to the tumor) with up to eight 2-week cycles of modified FOLFIRINOX chemotherapy.

ACT treatment will be given on Day 1 of each cycle of chemotherapy. Patients' well-being and side effects will be assessed at the same visits. The objective efficacy of the treatment will be assessed by CT scans every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Not deemed suitable for primary curative surgery and have radiographic and pathological disease consistent with inoperable LAPC or borderline resectable pancreatic cancer.
* Suitable to receive treatment with mFOLFIRINOX according to the Investigator's assessment.

Exclusion Criteria:

• Any prior anti-cancer treatment for pancreatic cancer (e.g. chemotherapy, surgery, radiation). Palliative bypass procedure and bile duct stenting are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
ORR (Overall response rate), defined as the number of participants with measurable disease at baseline who have a confirmed Complete Response or confirmed Partial Response according to RECIST Version 1.1. | From baseline to end of treatment (up to Week 24)

SECONDARY OUTCOMES:
Overall summary of TEAEs including number and percentage of participants with at least one TEAE. TEAEs will be summarized by System Organ Class and Preferred Term. TEAEs will be summarized by severity and causality. | From enrollment up to week 24
Change in maximum tumor diameter and volume summarized as the largest or the smallest percentage change from baseline. Independent central image review based on RECIST 1.1 criteria will be the primary analysis. | From baseline up to week 24
Median OS and proportion of participants alive at 6 months. | from baseline to week 24
The proportion of participants becoming eligible for resection as determined by local multidisciplinary team review | from baseline to week 24

CONTACTS AND LOCATIONS:
Locations (10):
- United States (7):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Stanford Cancer Center Palo Alto, Stanford, California
  - Beth Israel Deaconess Medical Center - Division of Hematology/Oncology, Boston, Massachusetts
  - Henry Ford Centre, Detroit, Michigan
  - Sidney Kimmel Cancer Center, Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Brown University Cancer Institute, Providence, Rhode Island
- United Kingdom (3):
  - CAMBRIDGE CANCER TRIALS CENTRE-Addenbrooke's Hospital, Cambridge, Cambridge
  - Gary Weston Centre- Imperial College Healthcare- Du Cane Road, Hammersmith, London
  - The Royal Marsden- Downs Road, Sutton, Surrey

IPD SHARING:
Plan to Share IPD: No